CLINICAL TRIAL: NCT02712944
Title: Effect of Testosterone Replacement on Erythropoietin Stimulating Agent Use in End Stage Renal Disease Patients
Brief Title: Testosterone Replacement in Renal Failure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped for procedural difficulties and lack of personnel
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L16-079
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone (Active Comparator): Testosterone intramuscular every 2 weeks
  Interventions: Drug: Testosterone
- Saline (Placebo Comparator): Saline intramuscular every 2 weeks
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Testosterone — Testosterone
  Arms: Testosterone
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
The purpose of this trial is to evaluate the effect of testosterone replacement in men with renal failure (on dialysis) who also have low testosterone. Specifically, the investigators will assess the change in requirement of Erythropoietin Stimulating agents.

DETAILED DESCRIPTION:
Testosterone replacement can increase hemoglobin count. This can therefore decrease the requirement of Erythropoietin Stimulating agents.

ELIGIBILITY:
Inclusion Criteria:

1. Men between ages of 18-80 years of age.
2. Renal failure on hemodialysis
3. Free testosterone <5 ng/dl.
4. Willing to be randomized to intramuscular (IM) testosterone or placebo
5. Currently getting intravenous Epoetin alfa

Exclusion Criteria:

1. Use of testosterone treatment currently or in the past 6 months, including use of over the counter androgen containing health supplements.
2. Congestive heart Failure, class III or IV.
3. Baseline hemoglobin of > 12 g/dl.
4. Allergic reactions to testosterone Vehicle (i.e. Peanut oil)
5. prostate specific antigen>4 ng/ml.
6. History of Prostate Cancer.
7. Liver enzymes >twice the upper limit of normal.
8. HIV or hepatitis C.
9. Severe untreated obstructive sleep apnea (defined as apnea-hypopnea index> 30).
10. Subjects on warfarin or other blood thinners.
11. Active infection (such as foot ulcer)
12. History of adverse events with testosterone use in past.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in dosage of Erythropoietin stimulating agents (ESA) | primary outcome will be measured at months 5 and 6.
  Comparison of dose of ESA in the 2 months prior to the start of the drug and in months 5 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MD, Principal Investigator — TTUHSC
Locations (1):
- TTUHSC-Permian Basin, Odessa, Texas, United States

IPD SHARING:
Plan to Share IPD: No